CLINICAL TRIAL: NCT04410666
Title: Antibacterial Effect of the Infusion of Green Tea (Camellia Sinensis) as a Mouthwash on Saliva and Bacterial Plaque
Brief Title: Antibacterial Effect of the Infusion of Green Tea Used as a Mouthwash on Saliva and Bacterial Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julieta María Méndez Romero (Other)
Responsible Party: Sponsor-Investigator, Julieta María Méndez Romero, Head of Writting and Publication Department, Regional Health Research Institute, Universidad Nacional de Caaguazu
Organization: Universidad Nacional de Caaguazu (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00139
Record Dates: First submitted 2020-05-24; First posted 2020-06-01 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Dental Plaque
Keywords: Saliva; Mouthwash; Green Tea; Oral bacteria
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: Experimental group: an infusion at 13%, with 13 g of green tea (commercially divided) in 100 ml of saline solution, at a temperature of approximately 90 ° C.
  Control group: distilled water, in sterile glass containers. Each application was 10 ml. applied for 1 minute.
Who Masked: Participant
Masking Description: It was single blind, since the patient did not wat treatment was receiving. It was used a placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GREEN TEA MOUTH WASH (Experimental): an infusion at 13%, with 13 g of green tea (commercially divided) in 100 ml of saline solution, at a temperature of approximately 90 ° C.
  Interventions: Other: Green Tea mouthwash
- Placebo (Placebo Comparator): distilled water, in sterile glass containers.
  Interventions: Other: Placebo Mouthwash

INTERVENTIONS:
Other: Green Tea mouthwash — an infusion at 13%, with 13 g of green tea (commercially divided) in 100 ml of saline solution, at a temperature of approximately 90 ° C, in sterile glass containers.
  Each application was 10 ml. applied for 1 minute.
  Arms: GREEN TEA MOUTH WASH
Other: Placebo Mouthwash — distilled water
  Arms: Placebo

SUMMARY:
Given that the participation of oral microorganisms in the development of the most prevalent pathologies of the oral cavity is unquestionable, efforts have been made to create agents that allow controlling these bacteria. The objective of this work was to analyze the antibacterial effect of green tea infusion used as a mouthwash on saliva and bacterial plaque. The green tea infusion was prepared at 13% at approximately 90 ° C, being the same applied to 14 participants from the 1st to the 5th grade (experimental group); and to other 14 participants the placebo was applied (control group). The antibacterial effect was determined by counting the colony forming units (CFU) in the cultures of samples of bacterial plaque and saliva, taken before the application of the infusion and immediately after.

DETAILED DESCRIPTION:
Oral diseases, including dental caries, is one of the most prevalent in the population. It is multifactorial and originates from the formation of the bacterial plaque and its non-elimination by physical and chemical hygiene methods.

The use of chemical agents to aid in the control of Bacterial Plaque has been the subject of study in many investigations. Today there is a variety of elements that can be use to carry out proper oral hygiene, such as toothbrushes, toothpastes, dental floss and mouthwash, all of them in a wide variety.

Often the lack of accessibility to these means problems in the hygiene in the population, either due to the lack of knowledge or the cost of obtaining them.

Therefore, the objective of analyzing the antibacterial effect of the infusion of green tea (camellia sinensis) used as a mouthwash on saliva and bacterial plaque was presented. The proposed research topic is relevant, since if green tea (camellia sinensis) is found to produce positive effects on bacterial plaque, it would serve to prevent its formation, thus helping to improve dental hygiene with an easy acquisition product and lower cost compared to other mouthwashes offered in the market, constituting a natural mouthwash.

ELIGIBILITY:
Inclusion Criteria:

* Participants that signed the informed consent

Exclusion Criteria:

* allergic to green tea (Camellia sinensis)
* ongoing medical or dental treatment that could interfere with the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08-21 (Actual); Primary Completion 2016-09-21 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
Bacterial plaque Stage 1 (Before intervention) | thorough study completion, an average of 24 hours
  The measure was done with the count of Colony forming units
Bacterial plaque Stage 2 (After intervention) | 1 minute after mouthwash use
  The measure was done with the count of Colony forming units
Antimicrobial effect | up to 24 hours, thorough study completion
  The measure was done with the difference in count of Colony forming units before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jazmin Servin, Principal Investigator — Facultad de Odontologia, Universidad Nacional de Caaguazu; Nelson Portillo, Study Director — Facultad de Odontologia, Universidad Nacional de Caaguazu
Locations (1):
- Facultad de Odontología, Universidad nacional de Caaguazu, Coronel Oviedo, Caaguazú Department, Paraguay

IPD SHARING:
Plan to Share IPD: Yes
By email
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From the time the protocol is available in clinical trials.gov and with no limit of time
Access Criteria: Researchers that want to know about the study and use the protocol

REFERENCES:
- [Background] Ardakani MR, Golmohammadi S, Ayremlou S, Taheri S, Daneshvar S, Meimandi M. Antibacterial effect of Iranian green-tea-containing mouthrinse vs chlorhexidine 0.2%: an in vitro study. Oral Health Prev Dent. 2014;12(2):157-62. doi: 10.3290/j.ohpd.a31663. PMID 24624389
- [Background] Megalaa N, Thirumurugan K, Kayalvizhi G, Sajeev R, Kayalvizhi EB, Ramesh V, Vargeese A. A comparative evaluation of the anticaries efficacy of herbal extracts (Tulsi and Black myrobalans) and sodium fluoride as mouthrinses in children: A randomized controlled trial. Indian J Dent Res. 2018 Nov-Dec;29(6):760-767. doi: 10.4103/ijdr.IJDR_790_16. PMID 30589005
- [Background] Ronanki S, Kulkarni S, Hemalatha R, Kumar M, Reddy P. Efficacy of commercially available chlorhexidine mouthrinses against specific oral microflora. Indian J Dent Res. 2016 Jan-Feb;27(1):48-53. doi: 10.4103/0970-9290.179816. PMID 27054861
- [Background] Hajiahmadi M, Yegdaneh A, Homayoni A, Parishani H, Moshkelgosha H, Salari-Moghaddam R. Comparative Evaluation of Efficacy of "Green Tea" and "Green Tea with Xylitol" Mouthwashes on the Salivary Streptococcus mutans and Lactobacillus Colony Count in Children: A Randomized Clinical Trial. J Contemp Dent Pract. 2019 Oct 1;20(10):1190-1194. PMID 31883255
- [Derived] Servin J, Mendez J, Portillo N, Villasanti U. Antibacterial effect of green tea infusion used as a mouthwash on saliva and bacterial plaque: a randomized controlled trial. Gen Dent. 2021 Sep-Oct;69(5):72-74. PMID 34424217